CLINICAL TRIAL: NCT07257731
Title: The Effect of Reformer Pilates Exercises on Functional Capacity, Balance, Muscular Endurance, and Quality of Life in Sedentary Women: A Randomized Controlled Trial
Brief Title: The Effect of Reformer Pilates on Functional Capacity, Balance, and Quality of Life in Sedentary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, ece turak, Principal Investigator and Physical Therapist (PT), Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 126/2025; IRB Protocol Number (Other: Istanbul Aydin University)
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sedentary Lifestyle; Functional Capacity
Keywords: Reduced Functional Capacity; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer Pilates Exercise Group (Experimental): 8-Week Reformer Pilates Intervention
  Interventions: Behavioral: Reformer Pilates Exercise Program
- Control Group (No Intervention): Usual Lifestyle

INTERVENTIONS:
Behavioral: Reformer Pilates Exercise Program — The Reformer Pilates Exercise Program was delivered over an 8-week period, consisting of 2 supervised sessions per week. Each session lasted 50 minutes and was administered by the same licensed Physical Therapist (PT) at the FLC Konsept Healthy Living Center. The exercises utilized the Reformer apparatus. The program was standardized but individually tailored by adjusting the spring resistance based on the participant's tolerance level and physical condition to ensure safe and effective exercise progression. The intervention focused on the six core principles of Pilates, targeting core stabilization, muscle strength, muscular endurance, flexibility, and balance to improve the overall physical fitness of sedentary women.
  Arms: Reformer Pilates Exercise Group

SUMMARY:
The objective of this randomized controlled trial is to evaluate the effect of Reformer Pilates exercises on functional capacity, balance, muscular endurance, and quality of life in sedentary women.

A total of 57 sedentary women were randomly assigned to either the Intervention Group (N=30) or the Control Group (N=27). Participants in the intervention group underwent an 8-week Reformer Pilates exercise program, consisting of 2 sessions per week, 50 minutes each. The control group maintained their usual lifestyle without intervention. All participants' functional capacity (1-minute sit-to-stand), balance (Functional Reach Test), muscular endurance (30-second push-up and sit-up tests), and quality of life (SF-36) were measured at baseline and at the end of the 8-week period.

DETAILED DESCRIPTION:
In the modern world, technological advances and evolving lifestyles have led to a significant global public health concern: the sedentary lifestyle. Sedentary behavior is defined by low energy expenditure ($\le 1.5$ METs) during activities like sitting or lying down. This trend contributes to the rise of chronic diseases, including cardiovascular conditions, Type 2 diabetes, and musculoskeletal disorders, placing a substantial burden on health systems.Women are particularly vulnerable to decreased physical activity due to physiological factors (e.g., pregnancy, menopause) and sociocultural aspects. This physical inactivity is linked to reduced muscle mass, bone density, poor functional capacity, and increased risk of falls. Furthermore, sedentary behaviors adversely affect psychosocial well-being, contributing to increased depression, anxiety, and a reduced overall quality of life.The Reformer Pilates method, based on principles such as core stabilization, control, and breathing, is a comprehensive exercise approach aimed at improving strength, flexibility, posture, and balance. The Reformer apparatus, with its springs and movable carriage, provides adjustable resistance and support, making it an efficient and safe exercise option, particularly for sedentary individuals. While existing literature supports the benefits of Pilates, there is a distinct gap regarding the combined effects of Reformer Pilates (not Mat Pilates) on the crucial parameters of functional capacity, balance, muscular endurance, and quality of life within the sedentary female population, using a high-evidence-level randomized controlled trial (RCT) design. This study aims to address this critical scientific gap.STUDY OBJECTIVE AND DESIGNThe primary objective of this study is to evaluate the effect of an 8-week Reformer Pilates exercise program on the levels of functional capacity, balance, muscular endurance, and quality of life in sedentary women, compared to a control group.This investigation is designed as a Randomized Controlled Trial (RCT). A total of 57 sedentary women were randomly assigned to either the Intervention Group (N=30) or the Control Group (N=27).INTERVENTION PROTOCOLIntervention Group: Participants in this group underwent an 8-week Reformer Pilates exercise program. The program involved 2 sessions per week, with each session lasting 50 minutes. All sessions were administered by the same physical therapist at a dedicated center (FLC Konsept Sağlıklı Yaşam Merkezi). The exercise protocol was standardized but personalized: the spring resistance on the Reformer apparatus was adjusted based on the individual participant's physical condition and tolerance to maximize efficiency and safety.Control Group: Participants in this group maintained their usual lifestyle and daily routine throughout the 8-week study period, without receiving any structured exercise intervention.OUTCOME MEASURESAll participants underwent comprehensive assessments at baseline and at the end of the 8-week intervention period. Measurements were taken by the same blinded physical therapist to ensure reliability and minimize bias.The primary outcome and secondary outcomes are defined as follows:Functional Capacity: Measured using the 1-Minute Sit-to-Stand Test.Balance: Measured using the Functional Reach Test.Muscular Endurance: Measured using the 30-Second Push-Up Test and the 30-Second Sit-Up Test.Quality of Life: Measured using the Short Form-36 Health Survey (SF-36) scale.

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Meeting the definition of sedentary (no participation in any regular exercise program within the last 6 months).
* Having sufficient ability to understand and comply with the study procedures.
* No physical or mental condition that would hinder safe participation in the study.
* Voluntarily agreeing to participate in the study and signing the informed consent form.

Exclusion Criteria:

* Presence of any neurological disorder that prevents safe exercise participation.
* Having an active sports life or currently participating in regular sports activities.
* Presence of cardiovascular, pulmonary, or serious orthopedic problems that contraindicate exercise (e.g., medical restriction by a physician).
* Being pregnant or breastfeeding.
* Presence of any acute pain or inflammatory condition.
* Having a known contraindication for Pilates exercises.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female (Kadın)
Enrollment: 57 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Functional Capacity 1-Minute Sit-to-Stand Test | Baseline and End of 8-Week Intervention
  The 1-Minute Sit-to-Stand Test (1-MSTST) is a standardized, reliable, and valid field test designed to assess lower-body strength, muscular endurance, and functional mobility in various populations, including sedentary adults.
  Procedure: The participant is instructed to stand up fully from a standard chair and sit down as many times as possible within a one-minute period, without using their arms for support.
  Scoring: The total number of complete repetitions performed correctly within 60 seconds is recorded as the test score. A higher number of repetitions indicates superior functional capacity and strength, often correlated with better mobility and reduced fall risk.

SECONDARY OUTCOMES:
Balance Functional Reach Test | Baseline and End of 8-Week Intervention
  The Functional Reach Test (FRT) is a simple, single-measure clinical assessment designed to evaluate dynamic balance and postural stability by quantifying a participant's ability to intentionally displace their center of gravity forward.
  Procedure: The participant stands next to a wall-mounted ruler, with the arm extended forward at 90 degrees. They are instructed to reach as far forward as possible without moving their feet or touching the wall. The measure is the maximum distance (typically in centimeters) between the initial position of the third metacarpal head and the final reached position.
  Interpretation: A higher score (longer reach distance) indicates superior balance, better postural control, and is associated with a lower risk of falls. Conversely, a reduced reach distance is a reliable predictor of increased fall risk and poor functional mobility.
Muscular Endurance 30-Second Push-Up Test | Baseline and End of 8-Week Intervention
  30-Second Push-Up Test: Measures the endurance of the upper body muscles (chest, shoulders, and triceps). Participants perform maximum repetitions in 30 seconds, using a modified knee-supported position for women (if applicable to your protocol). Scoring: The total number of complete and correct repetitions performed within the 30-second period for this test is recorded. A higher score indicates superior upper body muscular endurance.
Quality of Life Short Form-36 Health Survey (SF-36) | Baseline and End of 8-Week Intervention
  The Short Form-36 Health Survey (SF-36) is a validated, standardized, and self-administered questionnaire measuring generic health status and health-related quality of life. It provides scores on eight distinct health domains:
  Physical Functioning (PF)
  Role Limitations due to Physical Health (RP)
  Bodily Pain (BP)
  General Health (GH)
  Vitality (VT)
  Social Functioning (SF)
  Role Limitations due to Emotional Problems (RE)
  Mental Health (MH)
  These eight scales are summarized into two key components: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores range from 0 (worst health) to 100 (best health).
Muscular Endurance 30-Second Sit-Up Test | Baseline and End of 8-Week Intervention
  30-Second Sit-Up Test: Measures the endurance of the core (abdominal) musculature. Participants perform maximum repetitions in 30 seconds, typically with the knees bent and feet held, touching the elbow to the thigh for each repetition. Scoring: The total number of complete and correct repetitions performed within the 30-second period for this test is recorded. A higher score indicates superior core muscular endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) that support the results of this study will be shared upon reasonable request to the corresponding author, following the publication of the final results. The data will be de-identified to protect participant privacy. Data will be made available for researchers who provide a methodologically sound proposal and sign a data access agreement. The types of data shared will include the full protocol, statistical analysis plan, and the raw dataset after anonymization.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the primary publication date 5 years after the primary publication date
Access Criteria: Access will be granted to qualified academic and research collaborators who submit a written, methodologically sound research proposal. Data will be shared only after ethical review and approval by the Institutional Review Board (IRB) of Istanbul Aydin University and upon the signing of a formal Data Access Agreement (DAA) with the corresponding author. Access will be provided to the anonymized Individual Participant Data (IPD), the full study protocol, the Statistical Analysis Plan (SAP), the Informed Consent Form (ICF), the Clinical Study Report (CSR), and analytic code for ethically approved and scientifically justifiable research purposes.